CLINICAL TRIAL: NCT01742819
Title: Detection of Glaucoma Progression Study With Macular OCT Imaging
Brief Title: Advanced Glaucoma Progression Study
Acronym: AGPS
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Kouros Nouri-Mahdavi, Assistant Professor of Ophthalmology, University of California, Los Angeles
Other Study IDs: IRB# 11-003602; 1K23EY022659-01 (NIH)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Primary Open Angle Glaucoma; Pseudoexfoliative Glaucoma; Chronic Angle Closure Glaucoma
Keywords: Glaucoma, Optical Coherence Tomography, Progression
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced glaucoma: Patients with MD < -6 or visual field loss within the central 10 degrees of the visual field.

SUMMARY:
Glaucoma is one of the leading causes of blindness in the world. The key to prevention of visual loss from glaucoma is early detection of the disease or its progression and timely treatment. The proposed study will investigate the role of various tests in improving detection of disease progression in advanced glaucoma. Evaluation of the peripheral field of vision (visual field examination) remains the current standard for detection of progression in glaucoma. However, there is a lot of variability or inconsistency in eyes with advanced glaucoma, which could make it difficult to detect worsening of glaucoma with visual fields. The optic nerve demonstrates significant damage in such eyes and hence oftentimes repeat imaging of the optic nerve head is not helpful for detection of change. Therefore, imaging of the central retina (the innermost sensitive tissue lining the inside of the eye), called macula, has been proposed to supplant imaging of the nerve in eyes with severe glaucoma. The macula aids in detailed central vision. Since the macular retinal neural cells are the last ones to be affected in glaucoma, measurement of macular retinal thickness could provide significant information with regard to the course of glaucoma. In the proposed study, glaucoma patients will be tested and followed with various measurements done with newer versions of optical coherence tomography (OCT) imaging and visual field machines. The patients will undergo repeat imaging and visual field testing every 6 months over the course of 5 years. Rates of change will be estimated. We will explore if changes in various outcome measures derived from imaging are correlated with the corresponding visual field changes in glaucoma, and whether the former can be used as an alternative method for detecting simultaneous or subsequent glaucoma progression. The hypothesis for this proposed research is that macular OCT parameters are valid structural measures that can be used especially in advanced disease to follow the course of glaucoma.

DETAILED DESCRIPTION:
Glaucoma is a major public health issue worldwide and manifests clinically as a chronic progressive optic neuropathy with concomitant visual field (VF) loss. Glaucoma can cause significant visual disability and decreased quality of life (1). Based on WHO's report in 2002, glaucoma is the second cause of blindness. The key to prevention of visual loss from glaucoma is early detection of the disease or its progression and timely treatment. Glaucoma can be quite advanced at the time of initial detection. The prevalence of advanced glaucoma at the time of diagnosis varies but can be quite high. For example, the average VF mean deviation (MD) in patients diagnosed with glaucoma in the Los Angeles Latino Eye Study was -9.6 dB (2), which represents moderately advanced to severe glaucoma. Detection of progression in advanced stages of glaucoma continues to be challenging. Visual field examination remains the gold standard for detection of progression in advanced glaucoma. However, long-term VF variability or noise in such eyes is significant, which could confound detection of change. The optic nerve head and peripapillary retinal nerve fiber layer (RNFL) demonstrate significant damage in such eyes and hence are not helpful for detection of change. About 50% of retinal ganglion cells (RGCs) are located within 4-5 mm of the macular center (3). Since the macular RGCs are the last ones to be affected in glaucoma, measurement of macular retinal thickness or retinal sublayers could provide significant information with regard to the course of advanced glaucoma.

The macular retinal sublayers can now be measured with reasonable accuracy with SD- OCTs. There is some evidence that measurement of the macular ganglion cell complex (GCC, combined thickness of RNFL, RGC and inner plexiform layer or IPL), or macular retinal thickness or volume may detect early glaucoma with a performance that approximates that of circumpapillary RNFL thickness measurements (4,5). In addition, such macular measurements have proved to be very reproducible (4,6). Given this excellent reproducibility, macular outcome measures would be the main candidates for following glaucoma eyes with advanced damage, in which the macular region is essentially the only retinal area with residual RGCs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary open angle glaucoma, pseudoexfoliative glaucoma, and angle closure glaucoma
* Visual field MD of -6dB or worse OR visual field loss involvement at at least two points within the central 10 degrees of the field

Exclusion Criteria:

* Patient not within the ages of 40-80 years old
* Visual acuity worse than 20/50 at baseline
* Spherical refraction worse than 8D and cylindrical refraction worse than 3D
* Significant retinal or neurological diseases including diabetic retinopathy or age-related macular degeneration

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced glaucoma patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Visual field progression | 5 years
  Worsening of the MD and/or increased visual field loss within the central 10 degrees of the field.
Worsening of OCT measurements | 5 Years
  Worsening of macular and retinal nerve fiber layer (RNFL) OCT measurements.

SECONDARY OUTCOMES:
Contrast sensitivity | 5 years
  Looking at any changes in contrast sensitivity using the Vector Vision CSV-1000 eye chart.

CONTACTS AND LOCATIONS:
Overall Officials: Kouros Nouri-Mahdavi, MD, MSc, Principal Investigator — Jules Stein Eye Institute, UCLA
Locations (1):
- UCLA Jules Stein Eye Institute, Los Angeles, California, United States

REFERENCES:
- [Background] McKean-Cowdin R, Wang Y, Wu J, Azen SP, Varma R; Los Angeles Latino Eye Study Group. Impact of visual field loss on health-related quality of life in glaucoma: the Los Angeles Latino Eye Study. Ophthalmology. 2008 Jun;115(6):941-948.e1. doi: 10.1016/j.ophtha.2007.08.037. Epub 2007 Nov 12. PMID 17997485
- [Background] Varma R, Ying-Lai M, Francis BA, Nguyen BB, Deneen J, Wilson MR, Azen SP; Los Angeles Latino Eye Study Group. Prevalence of open-angle glaucoma and ocular hypertension in Latinos: the Los Angeles Latino Eye Study. Ophthalmology. 2004 Aug;111(8):1439-48. doi: 10.1016/j.ophtha.2004.01.025. PMID 15288969
- [Background] Curcio CA, Allen KA. Topography of ganglion cells in human retina. J Comp Neurol. 1990 Oct 1;300(1):5-25. doi: 10.1002/cne.903000103. PMID 2229487
- [Background] Tan O, Chopra V, Lu AT, Schuman JS, Ishikawa H, Wollstein G, Varma R, Huang D. Detection of macular ganglion cell loss in glaucoma by Fourier-domain optical coherence tomography. Ophthalmology. 2009 Dec;116(12):2305-14.e1-2. doi: 10.1016/j.ophtha.2009.05.025. Epub 2009 Sep 10. PMID 19744726
- [Background] Mori S, Hangai M, Sakamoto A, Yoshimura N. Spectral-domain optical coherence tomography measurement of macular volume for diagnosing glaucoma. J Glaucoma. 2010 Oct-Nov;19(8):528-34. doi: 10.1097/IJG.0b013e3181ca7acf. PMID 20164794
- [Background] Mwanza JC, Oakley JD, Budenz DL, Chang RT, Knight OJ, Feuer WJ. Macular ganglion cell-inner plexiform layer: automated detection and thickness reproducibility with spectral domain-optical coherence tomography in glaucoma. Invest Ophthalmol Vis Sci. 2011 Oct 21;52(11):8323-9. doi: 10.1167/iovs.11-7962. PMID 21917932
- [Derived] Lee JW, Morales E, Sharifipour F, Amini N, Yu F, Afifi AA, Coleman AL, Caprioli J, Nouri-Mahdavi K. The relationship between central visual field sensitivity and macular ganglion cell/inner plexiform layer thickness in glaucoma. Br J Ophthalmol. 2017 Aug;101(8):1052-1058. doi: 10.1136/bjophthalmol-2016-309208. Epub 2017 Jan 11. PMID 28077369